CLINICAL TRIAL: NCT07114159
Title: An Open-label Clinical Trial to Evaluate the Long-term Safety and Efficacy of Sacral Nerve Stimulation in Patients With Ulcerative Colitis
Brief Title: Long-term Safety and Efficacy of Sacral Nerve Stimulation in Patients With Ulcerative Colitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20232100-extension
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sacral nerve stimulation (Experimental)
  Interventions: Device: Sacral nerve stimulation

INTERVENTIONS:
Device: Sacral nerve stimulation — Device: G132 system, Beijing PINS Medical Co., China Neuromodulation was performed according to the usual protocol

SUMMARY:
Although the incidence of inflammatory bowel disease is stable in North American and European countries, the incidence of inflammatory bowel disease is increasing in newly industrialized countries, especially in China. The treatment drugs for ulcerative colitis include 5-aminosalicylic acid (5-ASA), glucocorticoids, immunosuppressants, and biological agents. The aim of this clinical trial is to evaluate the long-term safety and efficacy of sacral nerve stimulation in patients with ulcerative colitis

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* ulcerative colitis diagnosed for at least 3 mouths.
* Mayo score 6-12, Mayo endoscopic score 2-3 points
* resistant to medical treatment

Exclusion Criteria:

* Treatment-naive ulcerative colitis (no previous treatment)
* Acute severe ulcerative colitis
* Currently taking any biologicals
* Previous surgical treatment or severe colitis at imminent risk of surgery
* infective colitis
* Other systemic diseases
* Pregnancy and lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08-02 (Actual); Primary Completion 2032-12-01 (Estimated); Study Completion 2032-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Mayo score | From baseline to 8 years
  The range of Mayo score is 0-12, and higher scores mean worse outcome

SECONDARY OUTCOMES:
Clinical remission | From baseline to 8 years
  overall mayo score ≤2 [and no individual subscore >1]
Clinical response | From baseline to 8 years
  defined as the reduction of baseline scores by ≥3 points
Change from baseline in the Truelove and Witts Severity Index | From baseline to 8 years
  Truelove and Witts Severity Index
Endoscopic remission | From baseline to 8 years
  defined as Mayo endoscopic score ≤ 1
Fecal calprotectin levels | From baseline to 8 years
  fecal sample
erythrocyte sedimentation rate levels | From baseline to 8 years
  blood sample
C reactive protein levels | From baseline to 8 years
  blood sample
Inflammatory Bowel Disease Questionnaire Score | From baseline to 8 years
  The range of Inflammatory Bowel Disease Questionnaire Score is 32-224, and higher scores mean worse outcome
Hospital Anxiety and Depression scale score | From baseline to 8 years
  The range of Hospital Anxiety and Depression scale score is 0-21, and higher scores mean worse outcome
Gut microbiota profile | From baseline to 8 years
  fecal sample
The Pittsburgh Sleep Quality Index | From baseline to 8 years
  higher scores mean worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No